CLINICAL TRIAL: NCT07371637
Title: Charge Your Brainzzz: Evaluation of an Integrated Approach to Improve Teenagers' Sleep Health
Brief Title: Charge Your Brainzzz: Evaluation of the Effectiveness and Implementation of an Integrated Approach to Improve Dutch Teenagers' Sleep Health
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Maartje van Stralen, Associate Professor, VU University of Amsterdam
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CYB3
Record Dates: First submitted 2025-09-25; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-09

CONDITIONS: Intervention Effectiveness; Implementation Research
Keywords: sleep; adolescent; healthy school; charge your brainzzz; evaluation

STUDY DESIGN:
Intervention Model Description: One group will receive the CYB intervention, while the other group will serve as a control group getting regular Dutch secondary school education
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Charge Your Brainzzz
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Charge Your Brainzzz — Charge Your Brainzzz is a comprehensive health promoting school approach intervention, designed to help Dutch secondary school students improve their sleep and sleep hygiene habits. It is based on the Health Promoting School framework and includes all its four pillars, i.e. (1) an education component, (2) a set of components that focus on involving students' (home) environment, a set of school policy changes related to school start times, schools' digital communication activities and schools' stimulation of daytime physical activity of students, and, lastly, (4) a set of tools that school health professionals can use to facilitate the early detection of potential (future) student sleep problems.
  Arms: Intervention group

SUMMARY:
Poor sleep among teenagers is a major public health issue. Studies show that in the Netherlands, nearly half of adolescents don't wake up feeling rested, one in five feel sleepy during the day, one in four regularly wake up at night, 65% rate their own sleep quality as poor, and 43% sleep less than the recommended 8-10 hours per night. Over the past decade, teenagers' average sleep time has dropped by about 40 minutes.

Good sleep health means having a regular sleep rhythm with about 8-10 hours of quality sleep each night. This is crucial, because poor sleep in teenagers can lead to problems with thinking, learning, concentration, and school performance. In the long run, it also increases the risk of serious health issues such as anxiety, depression, obesity, diabetes, cardiovascular disease, and even dementia.

Because of these risks, schools, municipalities, and public health services are calling for effective ways to prevent sleep problems among teenagers. The Dutch "Healthy School" program has recently added sleep as a core theme, but proven, practical interventions are still lacking.

To address this gap, the Charge Your Brainzzz (CYB) program was developed. CYB is a comprehensive approach designed to help secondary school students improve their sleep and mental well-being. It is based on the Healthy School framework and includes all four pillars: education, environment, policy, and early detection.

In 2024, a pilot study tested the CYB approach for its initial effectiveness and suitability. Early results showed positive changes in sleep outcomes and strong appreciation from both schools and students. However, before CYB can be rolled out nationwide, more evidence is needed on its effectiveness, fit with schools, and how it can be sustained over time.

That's why this project will conduct a large-scale evaluation of both the impact of CYB and the processes needed for successful implementation. Alongside the effectiveness study, a practical roadmap will be co-created with schools, Healthy School Advisors, and local coordinators to ensure that CYB can be optimally implemented, sustained, and scaled up across schools, municipalities, and public health services across the Dutch public health landscape.

DETAILED DESCRIPTION:
Poor sleep health among adolescents is a major public health problem. In the Netherlands, nearly half of adolescents report not waking up feeling rested, one in five say they feel sleepy during the day, one in four regularly do not sleep through the night, 65% rate their own sleep quality as poor, and 43% sleep less than the recommended 8-10 hours per night. Over the past ten years, adolescents' average sleep duration has decreased by about 40 minutes.

Sleep health refers to maintaining a regular sleep rhythm of approximately 8-10 hours of good-quality sleep per night. Sleep health is extremely important, because when teenagers sleep poorly, they may experience declines in cognition, learning ability, concentration, and school performance. Moreover, poor sleep in adolescence increases the risk of long-term health problems such as anxiety and depression, obesity, diabetes, cardiovascular disease, and dementia.

From both research and the practical experience of schools, municipalities, and public health services, there is a strong demand for effective interventions to address these problems through prevention among teenagers. The Dutch "Healthy School" program (Gezonde School) shares this sense of urgency and has recently added sleep as a core theme. However, proven effective interventions for practice are still lacking.

To fill this gap, the integrated Charge Your Brainzzz (CYB) approach was recently developed to support secondary school students in improving their sleep and mental well-being. The approach is based on the Healthy School framework, with well-substantiated applications of all four Healthy School pillars: Education, Environment, Policy, and Early Detection.

In 2024, a pilot study was conducted to evaluate the initial effectiveness and suitability of the CYB approach (Pilot Study results in draft, 2025). Preliminary results from this pilot evaluation showed positive changes in sleep outcomes and strong appreciation from both schools and adolescents. However, before schools, municipalities, and public health services can implement CYB nationwide within the Healthy School framework, it is important to establish clarity about the program's effectiveness, appropriateness, sustainability processes, and, above all, its efficacy. Therefore, a sufficiently large, controlled evaluation study is needed to assess both effectiveness in practice and the processes of implementation and sustainability.

This project will therefore evaluate both the effectiveness as well as the implementation and sustainability processes of the CYB approach. In parallel, a step-by-step plan will be co-created with schools, Healthy School Advisors, and local JOGG coordinators to enable them to implement, sustain, and scale up the CYB approach across schools, municipalities, and public health services.

ELIGIBILITY:
Inclusion Criteria:

* Dutch regular secondary schools that include at least one vocational track (VMBO)
* First-year students enrolled in the VMBO tracks of participating schools
* Teachers, school health professionals, school care coordinators, school management, and the regional municipal health service's (GGD) Healthy School advisors who work with at least one of the participating schools

Exclusion Criteria:

* non-regular Dutch secondary schools / special education

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Subjective sleep health | From the start of the intervention until 6 months after its completion
  Subjective sleep health will be assessed using a concise questionnaire that comprehensively covers the submeasures (1) sleep duration, (2) sleep quality, (3) sleep efficiency, (4) bedtime routines/sleep hygiene, (5) sleep timing, and (6) daytime sleepiness [1,2]. In addition to sleep health, the most relevant behavioral determinants will be measured at each assessment point, alongside the direct targets of the CYB program. These include, for example, the presence of household rules regarding bedtimes and wake-up times, as well as adolescents' sleep hygiene practices, with particular attention to evening screen use and the presence of a mobile phone in the bedroom at night.
  Time frame of data collection: prior to implementation of the program (T0), within two weeks after completion of the educational component, (T1), and at six-month follow-up after T1 (T2).
  1. Buysse (2014). https://doi.org/10.5665/sleep.3298
  2. Meltzer (2021). https://doi.org/10.1016/j.smrv.2021.101425
Objective sleep duration | During five weekdays directly prior to the start of the intervention's implementation, within two weeks after its completion, and six months thereafter.
  A random selection of approximately two classes per participating school will wear GeneActiv sleep monitors during the three measurement periods (T0, T1, T2) to objectively assess sleep duration and sleep quality. These sleep monitors will be worn continuously on the wrist for a period of five weekdays. These devices measure the activity pattern, temperature, and ambient light surrounding the student wearing them.
Objective sleep quality | During five weekdays directly prior to the start of the intervention's implementation, within two weeks after its completion, and six months thereafter.
  A random selection of approximately two classes per participating school will wear GeneActiv sleep monitors during the three measurement periods (T0, T1, T2) to objectively assess sleep duration and sleep quality. These sleep monitors will be worn continuously on the wrist for a period of five weekdays. These devices measure the activity pattern, temperature, and ambient light surrounding the student wearing them. Additionally, during these days, students will complete a sleep diary each morning (approximately 5 minutes).
Subjective Sleep Duration | During five weekdays directly prior to the start of the intervention's implementation, within two weeks after its completion, and six months thereafter.
  All participating students will complete a sleep diary each morning (approximately 5 minutes) in which they report their sleep duration.

SECONDARY OUTCOMES:
Students' knowledge on healthy sleep | Prior to intervention implementation (T0), within two weeks after intervention completion (T1), and six months after T1.
  An assessment of students' knowledge on healthy sleep, based on the content of what's being taught via the CYB intervention program
Students' attitude towards sleep health | Prior to intervention implementation (T0), within two weeks after intervention completion (T1), and six months after T1.
  An assessment of students' attitude towards healthy sleep and their awareness of its importance to their health, wellbeing and ability to learn, based on the content of what's being taught via the CYB intervention program
Students' self-efficacy in relation to their sleep health | Prior to intervention implementation (T0), within two weeks after intervention completion (T1), and six months after T1.
  An assessment of students' self-efficacy/skills in relation to regulating their healthy sleep habits, based on the content of what's being taught via the CYB intervention program
Students' subjective norms in relation to sleep health of their peers and parents | Prior to intervention implementation (T0), within two weeks after intervention completion (T1), and six months after T1.
  An assessment of the subjective norm that students experience in their social environment in relation to healthy sleep habits.
Students' behavioral intention to sleep healthier | Prior to intervention implementation (T0), within two weeks after intervention completion (T1), and six months after T1.
  An assessment of whether students have the intention to exhibit healthier sleep habitss as a consequence of their school participating in the CYB intervention program
Students' sleep hygiene practices | Prior to intervention implementation (T0), within two weeks after intervention completion (T1), and six months after T1.
  An assessment of students' pre-sleep habits, or sleep hygiene practices, based on the content of what's being taught via the CYB intervention program
Appreciation and acceptance of the intervention | In the first school year following the start of the implementation of the program (T1), and again six months later (T2)
  In the first school year following the start of the implementation of the program (T1), and again six months later (T2), semi-structured interviews will be conducted with implementers of the CYB approach, i.e., the various school professionals involved, in order to monitor and evaluate the implementation within the school setting
Facilitators and barriers in relation to the intervention's adoption, implementation and sustainment | In the first school year following the start of the implementation of the program (T1), and again six months later (T2)
  An assessment of the facilitators and barriers in relation to the adoption, implementation and sustainment processes of the CYB program
Ripple effects mapping | Every 4 months after the start of the intervention's implementation
  The broader impact of the CYB program will be evaluated using the innovative systems-based evaluation method Ripple Effects Mapping (REM). Through this approach, we will work with implementers of the CYB program to capture, in real time, the overall impact of CYB. Ripple Effects Mapping provides an overview of both the direct and indirect effects of the various program components. These may occur within schools, within municipalities, at the level of the CYB program owner, or in other ways in which the intervention may have had unforeseen impact.
  REM sessions will commence once the CYB program has been expanded with activities beyond the school setting and will subsequently take place approximately every four months. During these sessions, time will be devoted to reviewing the actions and changes that have occurred in the past four months (retrospective analysis) as well as those that are expected or planned for the coming four months.

CONTACTS AND LOCATIONS:
Overall Officials: Maartje M van Stralen, PhD, Principal Investigator — VU University of Amsterdam
Locations (1):
- VU University, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: intervention description — https://chargeyourbrainzzz.nl/